CLINICAL TRIAL: NCT04964466
Title: Growth Factor Availability and Release Kinetics in PRF Versus GEM21S With and Without Bone Substitutes: An In Vitro Analysis
Brief Title: Release Kinetics in PRF Versus GEM21S With and Without Bone Substitutes: An In Vitro Analysis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria L. Geisinger, DDS, MS, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300005971; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Bone Loss
Keywords: Platelet concentrates; Platelet-rich fibrin; Growth factor; Bone morphogenic protein
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Prolactin-Releasing Hormone; Bone Substitutes; Becaplermin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood will be harvested to form PRF matrices, which will be used in Vitro clinical assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Amount of PDGF-BB in PRF preparation vs. GEM21: The release kinetics of PDGF-BB will be assessed for one PRF preparation from each of the six individual participants and one GEM 21S sample. The quantification will be performed at 60 minutes, 8 hours, 1 day, 3 days, and 10 days. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Interventions: Biological: Amount of PDGF-BB in PRF preparation vs. GEM21
- PDGF-BB available in PRF + bone substitutes vs. rhPDGF-BB+ bone substitutes: Growth factor release assessments will be made to determine the PDGF-BB present in the six prepared samples of the following: 1) PRF + mineralized freeze-dried corticocancellous allograft, 2) PRF + xenograft, and 3) PRF + B-TCP. Assessments will also be made for one sample of each of the following: 1) rhPDGF-BB + freeze-dried bone allograft, 2) rhPDGF-BB + xenograft, and 3) rhPDGF-BB+ B-TCP preparation. This assessment will be made at 60 minutes following the incorporation of the bone graft materials. During this time period, the samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At 60 minutes after preparation, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Interventions: Biological: Amount of PDGF-BB available in PRF + bone substitutes vs. rhPDGF-BB+ bone substitutes following preparation
- : Release kinetics of PDGF-BB in PRF + bone substitutes vs. rhPDGF-BB + bone substitutes: The release kinetics of PDGF-BB will be assessed for six preparations of each of following: 1) PRF+ mineralized freeze-dried corticocancellous allograft, 2) PRF + bone xenograft, and 3) PRF + B-TCP. The release kinetics of PDGF-BB will also be assessed for one preparations of each of following: 1) rhPDGF-BB + mineralized freeze-dried corticocancellous allograft, 2) rhPDGF-BB + bone xenograft, 3) rhPDGF-BB + TCP. The quantification will be performed at 60 minutes, 8 hours, 1 day, 3 days, and 10 days. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Interventions: Biological: Release kinetics of PDGF-BB in PRF + bone substitutes vs. rhPDGF-BB + bone substitutes
- Release kinetics of PDGF-BB in rhPDGF-BB + PRF + bone substitutes: The quantification will be performed at 60 minutes, 8 hours, 1 day, 3 days, and 10 days. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Interventions: Biological: Release kinetics of PDGF-BB in rhPDGF-BB + PRF + bone substitutes

INTERVENTIONS:
Biological: Amount of PDGF-BB in PRF preparation vs. GEM21 — The quantification will be performed at 60 minutes, 8 hours, 1 day, 3 days, and 10 days. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Groups: Amount of PDGF-BB in PRF preparation vs. GEM21
Biological: Amount of PDGF-BB available in PRF + bone substitutes vs. rhPDGF-BB+ bone substitutes following preparation — Growth factor release assessments will be made to determine the PDGF-BB present in the six prepared samples of the following: 1) PRF + mineralized freeze-dried corticocancellous allograft, 2) PRF + xenograft, and 3) PRF + B-TCP. Assessments will also be made for one sample of each of the following: 1) rhPDGF-BB + freeze-dried bone allograft, 2) rhPDGF-BB + xenograft, and 3) rhPDGF-BB+ B-TCP preparation. This assessment will be made at 60 minutes following the incorporation of the bone graft materials. During this time period, the samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At 60 minutes after preparation, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Groups: PDGF-BB available in PRF + bone substitutes vs. rhPDGF-BB+ bone substitutes
Biological: Release kinetics of PDGF-BB in PRF + bone substitutes vs. rhPDGF-BB + bone substitutes — The release kinetics of PDGF-BB will be assessed for six preparations of each of following: 1) PRF+ mineralized freeze-dried corticocancellous allograft, 2) PRF + bone xenograft, and 3) PRF + B-TCP. The release kinetics of PDGF-BB will also be assessed for one preparations of each of following: 1) rhPDGF-BB + mineralized freeze-dried corticocancellous allograft, 2) rhPDGF-BB + bone xenograft, 3) rhPDGF-BB + TCP. The quantification will be performed at 60 minutes, 8 hours, 1 day, 3 days, and 10 days. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Groups: : Release kinetics of PDGF-BB in PRF + bone substitutes vs. rhPDGF-BB + bone substitutes
Biological: Release kinetics of PDGF-BB in rhPDGF-BB + PRF + bone substitutes — The quantification will be performed at 60 minutes, 8 hours, 1 day, 3 days, and 10 days. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol. The samples will each be placed in a cell incubator at 37°C to allow for growth factor release into a phosphate-buffered saline. At each desired time point assessment, 2 ml of the sample will be collected, frozen, and replaced with 2 ml of additional phosphate-buffered saline. The protein quantification will be carried out using ELISA assay according to manufacturer's protocol.
  Groups: Release kinetics of PDGF-BB in rhPDGF-BB + PRF + bone substitutes

SUMMARY:
This study is seeking to evaluate that platelet-derived growth factor-BB (PDGF-BB) is a proven wound healing and osteogenic protein that plays a critical role in wound healing and previous research has demonstrated a non-linear response where higher dosages produced less effect. As Platelet Rich Fibrin (PRF) contains numerous platelets, it contains PDGF-BB, but at levels lower than in the commercially available product and with inter-individual variation, GEM21S. To achieve both ideal handling and achieve ideal levels of PDGF-BB, there is a rationale to add GEM 21S recombinant human platelet-derived growth factor-BB (rhPDGF) to a bone graft prior to making "sticky bone".

DETAILED DESCRIPTION:
Innovations in biomedicine and recombinant protein technology show promising advances for the regeneration of advanced alveolar defects. Recombinant growth factors and biologics encourage minimally invasive procedures with improved clinical outcomes/healing times in complex oral surgery procedures. PDGF-BB is a growth factor that is known to be a potent mitogen and chemotactic agent for cells important in wound healing and bone regeneration. PDGF-BB is also a strong angiogenic agent. These properties provide a solid biological mechanism of action and rationale for the widespread use of rhPDGF-BB in dental and orthopedic surgery, as well as in the treatment of difficult soft tissue wounds. Practically, two sources of supra-physiologic levels PDGF-BB are currently available for use in dental hard and soft tissue defects: 1) Platelet concentrates (PRF/PRF); and 2) GEM 21S, which contains recombinant human PDGF-BB (rhPDGF-BB). Platelet rich plasma was first introduced to dentistry in 1998 by Robert Marx. Since then, other autologous products have evolved. Platelet rich fibrin (PRF) is one that is used daily in various clinical scenarios, including guided bone regeneration. The rationale for its use is due to the supraphysiologic concentration of growth factors (ie PDGF-BB) and cells to enhance would healing. Clinicians also frequently incorporate PRF to bone grating materials to improve handling properties of the graft material, also referred to as "sticky bone". However, the literature varies greatly on the believed mechanism of action and the therapeutic benefits claimed by their supporters. The rationale for this proposed study that PDGF-BB is a proven wound healing and osteogenic protein, but there are clinically insignificant amounts of PDGF-BB in PRF. Therefore, there is a rationale to add GEM 21S (rhPDGF) to a bone graft prior to making "sticky bone" with PRF. This would provide clinicians the benefits of a clinically proven and consistent dose of rhPDGF to improve wound healing and bone formation in conjunction with the benefits of the improved handling (i.e. sticky bone) from the addition of the PRF.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Able to read and understand informed consent document
* Systemically healthy, non-smoker, no medications

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting healing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must be at least 18 years old with demonstrated ability to understand and consent to the proposed study procedures. Subjects treated in the UAB School of Dentistry Periodontal Clinic and scheduled for procedures using platelet rich fibrin (PRF) were performed.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To quantify any difference in the release of PDGF-BB after application to rhPDGF-BB and PRF | From baseline to 10 days
  The quantities of PDGF-BB statistical analysis using a two-way analysis of variance for the proliferation assay with Bonferroni test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States